CLINICAL TRIAL: NCT02439242
Title: Correlation Between the Pulse Pressure / Heart Rate Ratio Variations and Stroke Volume Variations During Fluid Challenge.
Brief Title: Correlation Between ΔPP/HR and ΔSV During Fluid Challenge.
Acronym: ΔPP/HRvsΔSV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: ΔPP/HR vs ΔSV
Record Dates: First submitted 2015-04-02; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Hypovolemia
Keywords: stroke volume, haemodynamic, fluid resucitation
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fluid challenge of saline — 250 ml of saline
  Other Names: ΔPP/HR and ΔSV

SUMMARY:
In high perioperative risk patients, guidelines suggest intraoperative haemodynamic optimization by measurement of stroke volume (SV) to guide fluid resucitation.This strategy requires an invasive monitoring and learning. Some studies tried to find SV surrogates based on haemodynamic usual parameters. In an experimental hemorrhagic shock, SV was correlated to the pulse pressure (PP) / heart rate (HR) ratio.

The investigators hypothesized that SV variations (ΔSV) would be correlated to the PP/HR ratio variations (ΔPP / HR) during fluid challenge, and ΔPP / HR would be able to detect a ΔSV greater than 10%.

ELIGIBILITY:
Inclusion Criteria:

* a suspected hypovolemia, based on clinical or paraclinical parameters.
* a fluid challenge decision at the discretion of the anaesthesiologist physician in charge of the patient.

Exclusion Criteria:

* Minor or major patient under guardianship,
* oesophageal Diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General anaesthesia.Orotracheal intubation and mechanical ventilation Advanced Haemodynamic Monitoring intraoperative ( arterial pressure catheter, oesophageal Doppler)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
correlation by linear regression between variations of the ratio PP/HR ( in percentage) and variations of SV ( in percentage) during fluid challenge | 18 months

SECONDARY OUTCOMES:
Area under the receiver operating characteristic curve (AUC roc) of the ability of variations of the ratio PP/HR ( in percentage)during fluid challenge to predict an increase of SV greater than 10% | 18 month

CONTACTS AND LOCATIONS:
Overall Officials: Olivier REBET, Principal Investigator — CHU CAEN
Locations (1):
- CAEN University Hospital, Caen, Basse Normandie, France